CLINICAL TRIAL: NCT00236938
Title: Efficacy and Safety of Venofer (Iron Sucrose Injection USP) in Patients Receiving Peritoneal Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VEN02021 / 1VEN02022
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Results first posted 2009-09-07 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Anemia
Keywords: iron; peritoneal dialysis; anemia
MeSH Terms: conditions — Anemia | interventions — Ferric Oxide, Saccharated; Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Fixed dose of erythropoietin (EPO) and Venofer (300mg) administered intravenous infusion over 1.5 hours on Days 1 and 15, and Venofer (400mg) administered intravenous infusion over 2.5 hours on Day 29.
  Interventions: Drug: Venofer and stable erythropoietin (EPO) regimen
- Group B (Active Comparator): Stable erythropoietin (EPO) dose and no supplemental iron.
  Interventions: Drug: stable erythropoietin (EPO) regimen

INTERVENTIONS:
Drug: Venofer and stable erythropoietin (EPO) regimen — Fixed dose of erythropoietin (EPO) and Venofer (300mg) administered intravenous infusion over 1.5 hours on Days 1 and 15, and Venofer (400mg) administered intravenous infusion over 2.5 hours on Day 29.
  Other Names: Iron Sucrose
  Arms: Group A
Drug: stable erythropoietin (EPO) regimen — Stable erythropoietin (EPO) dose and no supplemental iron.
  Other Names: EPO
  Arms: Group B

SUMMARY:
This is a open-label, prospective study comparing intravenous (IV) iron supplementation to standard care in anemic patents undergoing peritoneal dialysis.

DETAILED DESCRIPTION:
This is an open-label, prospective study comparing IV iron supplementation to standard care in anemic patients undergoing peritoneal dialysis. After successfully completing a 6 month enrollment period, qualifying patients were randomized to receive 1000mg of IV iron over a four week period, or no iron supplementation. Erythropoietin regimen was to remain stable. Patients were followed to day 71 for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin >= 9.5 and <= 11.5 g/dL.
* Ferritin <= 500 ng/ml.
* Serum Transferrin Saturation (TSAT) <= 25%.
* Stable erythropoietin (EPO) Regimen for 8 weeks.
* No iron for last 4 weeks before randomization.

Exclusion Criteria:

* Known Sensitivity to Iron Sucrose.
* Suffering concomitant severe diseases of the liver & cardiovascular system.
* Pregnancy / Lactation.
* Inadequate dialysis.
* Current treatment for asthma.
* Significant blood loss.
* Probability of need for transfusion or transfusion within 1 week of enrollment.
* Anticipated major surgery.
* Hemochromatosis / hemosiderosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2002-07; Primary Completion 2004-09 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Falone, MD, Study Director — American Regent, Inc.

REFERENCES:
- [Background] Singh H, Reed J, Noble S, Cangiano JL, Van Wyck DB; United States Iron Sucrose (Venofer) Clinical Trials Group. Effect of intravenous iron sucrose in peritoneal dialysis patients who receive erythropoiesis-stimulating agents for anemia: a randomized, controlled trial. Clin J Am Soc Nephrol. 2006 May;1(3):475-82. doi: 10.2215/CJN.01541005. Epub 2006 Mar 29. PMID 17699248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 29, 2002 - September 6, 2004 Locations: Hospitals and Medical Clinics
Groups:
- Group A: Venofer and Erythropoietin EPO Fixed Dose: Fixed dose of erythropoietin (EPO) and Venofer (300mg) administered intravenous infusion over 1.5 hours on Days 1 and 15, and Venofer (400mg) administered intravenous infusion over 2.5 hours on Day 29.
- Group B: Erythropoietin EPO Fixed Dose Only: Stable erythropoietin (EPO) dose and no supplemental iron.
Period: Overall Study
Arm/Group | Group A: Venofer and Erythropoietin EPO Fixed Dose | Group B: Erythropoietin EPO Fixed Dose Only
Started | 75 | 46
Completed | 62 | 26
Not Completed | 13 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Venofer and Erythropoietin EPO Fixed Dose | Group B: Erythropoietin EPO Fixed Dose Only | Total
Number analyzed (Participants) | 75 | 46 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 10 | 24
  >=65 years | 61 | 36 | 97
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 25 | 71
  Male | 29 | 21 | 50

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to the Highest Hemoglobin up to Day 71
Time Frame: Change from Baseline up to Day 71
Population: Intent-to-Treat Population (ITT): All safety population subjects who received at least 1 dose of study medication or EPO and had at least 1 post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Group A: Venofer and Erythropoietin EPO Fixed Dose | Group B: Erythropoietin EPO Fixed Dose Only
Number analyzed (Participants) | 66 | 30
g/dL | 1.3 (1.10) | .7 (1.10)

2. Secondary Outcome: The Mean Change From Baseline to the Highest Serum Transferrin Saturation (TSAT) up to Day 71
Time Frame: Change from Baseline up to Day 71
Population: Intent-to-Treat Population (ITT)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Group A: Venofer and Erythropoietin EPO Fixed Dose | Group B: Erythropoietin EPO Fixed Dose Only
Number analyzed (Participants) | 66 | 30
percentage of change | 18.176 (15.53) | 10.383 (12.27)

3. Secondary Outcome: The Mean Change From Baseline to the Highest Ferritin up to Day 71
Time Frame: Change from Baseline up to Day 71
Population: Intent-to-Treat Population (ITT)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A: Venofer and Erythropoietin EPO Fixed Dose | Group B: Erythropoietin EPO Fixed Dose Only
Number analyzed (Participants) | 66 | 30
ng/mL | 545.05 (585.8) | 70.523 (159.7)

4. Secondary Outcome: The Mean Change From Baseline to the Highest Reticulocyte Count up to Day 71
Time Frame: Change from Baseline up to Day 71
Population: Intent-to-Treat Population (ITT)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Group A: Venofer and Erythropoietin EPO Fixed Dose | Group B: Erythropoietin EPO Fixed Dose Only
Number analyzed (Participants) | 66 | 30
percentage of change | 0.7226 (1.36) | 0.4630 (1.01)

ADVERSE EVENTS:
Time Frame: 2 years and 2 months
Arm/Group | Group A: Venofer and Erythropoietin EPO Fixed Dose | Group B: Erythropoietin EPO Fixed Dose Only
Serious Adverse Events (participants affected / at risk) | 9/75 | 5/46
Other Adverse Events (participants affected / at risk) | 33/75 | 20/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Venofer and Erythropoietin EPO Fixed Dose (N=75) | Group B: Erythropoietin EPO Fixed Dose Only (N=46)
Anemia NOS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gangrene NOS (Vascular disorders) | 1 (1) | 0 (0)
Hyperglycemia NOS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension NOS (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Localized infection (Infections and infestations) | 0 (0) | 1 (1)
Lower limb fracture NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lymph node tuberculosis NOS (Infections and infestations) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Peritoneal infection (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory tract infection NOS (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Venofer and Erythropoietin EPO Fixed Dose (N=75) | Group B: Erythropoietin EPO Fixed Dose Only (N=46)
Abdominal pain NOS (Gastrointestinal disorders) | 3 (5) | 3 (3)
Catheter site infection (Infections and infestations) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diarrhea NOS (Gastrointestinal disorders) | 6 (9) | 2 (2)
Hypertension NOS (Vascular disorders) | 6 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (6) | 2 (2)
Oedema peripheral (General disorders) | 4 (6) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Peritoneal infection (Infections and infestations) | 4 (4) | 3 (3)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0)
Vomiting NOS (Gastrointestinal disorders) | 6 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less